CLINICAL TRIAL: NCT04479956
Title: Microwave Venous Ablation in Comparison to Radiofrequency Ablation, Laser Ablation and Surgical Ligation in Management of Great Saphenous Vein Incompetence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: R.20.06.905 - 2020/06/18
Record Dates: First submitted 2020-07-17; First posted 2020-07-21 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Varicose Veins
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Intervention Model Description: Randomized controlled Prospective study
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Computer Based
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Surgical Ligation (Experimental): Conventional surgical procedures will carried out through a 3-4 cm incision in the groin. The trunk of GSV and the tributaries will be ligated and divided.
  Interventions: Procedure: Varicose vein surgery
- Microwave group (Experimental): The microwave treating wire (Microwave Intracavity Coagulation System; Shanghai Medical Electronics, Shanghai, China) will be inserted into the GSV until it reached the medial aspect of ankle, guided by a light that illuminated the tip of the wire. Then, GSV will be ablated using pulse mode at 20-30 W. The treating wire will be withdrawn at 2-4 mm/s, with the ablation time lasting 2 s (energy delivery to the GSV was estimated at around 80 J/cm); the treatment parameters will be based on a previous report. Tumescence will be used in all patients with 0.9% saline containing 20 mL 2% lidocaine with 1: 200,000 adrenaline and 20 mL 0.5% levobupivacaine in 1 L 0.9% saline.
  Interventions: Procedure: Varicose vein surgery
- Laser ablation group (Experimental): Endovenous Laser Ablation (EVLA) uses a laser Fiber, which is inserted into the abnormal vein via a small skin puncture.using 1470 nm laser and a "radial" fiber for less discomfort. Two weeks later the "branch vessels" have reduced in size
  Interventions: Procedure: Varicose vein surgery
- Radiofrequency ablation group (Experimental): inserts a small catheter into the diseased vein through a small incision, using ultrasound guidance for an accurate and live view. Consistent and uniform heat is delivered to contract the collagen in the vein walls, causing them to collapse and close. After the vein is closed the treated vein is gradually absorbed into surrounding tissue.
  Interventions: Procedure: Varicose vein surgery

INTERVENTIONS:
Procedure: Varicose vein surgery — sapheno-femoral junction (SFJ) incompetence, GSV reflux from the groin to below the knee

SUMMARY:
The authors will aim to compare microwave therapy with other lines of management radio-frequency ablation, Laser ablation and surgical ligation; regarding time to recurrence rate, ulcer-free time, and health-related quality of life. In a randomized controlled study,The study will be conducted at the department of vascular surgery in Mansoura university hospitals

DETAILED DESCRIPTION:
INTRODUCTION:

Chronic venous disease (CVD) is one of the most common pathologies in the general population of adults in both industrialized and developing countries.1 the most severe form of CVD is venous ulceration with an overall prevalence of about 1 % in the adult population, which increases with age and is more common in women and obese patients. Venous ulcers significantly impair quality of life, and their treatment places a heavy financial burden upon healthcare systems. Varicose veins (VVS) is a common disease in adults, and VVS without skin changes are present in about 20% of the population, while active ulcers are found in 0.5%. The traditional surgical treatment of VVS is high ligation of the great saphenous vein (GSV), axial stripping and phlebotomy, but the postoperative clinical recurrence is as high as 60%.

Recently, minimally invasive techniques, such as endovenous laser ablation (EVLA) and radiofrequency ablation (RFA), have become widely used for the treatment of VVS. Several reports have shown Several reports have shown that endovenous techniques are as effective as traditional procedures.

Endovenous Microwave Ablation (EMA) for the treatment of VVS differs from the other endovenous methods, and no specific dose regime has been established for this system. Thus, it is unclear if EMA is more or less effective than conventional surgery, or whether it has any additional benefits. In this study, we compared the clinical outcome of high ligation and stripping (HLS) with EMA. Postoperative quality of life (QoL) analysis was assessed using the Aberdeen Varicose Vein Questionnaire (AVVQ) and Venous Clinical Severity Score (VCSS).

Aim of the work: Aimed to compare microwave therapy with other lines of management radiofrequency ablation, Laser ablation and surgical ligation; regarding time to recurrence rate, ulcer-free time, and health-related quality of life.

Patients and methods Study location: The study will be conducted at the department of vascular surgery in Mansoura university hospitals Type of study: Randomized controlled Prospective study Study duration: 2 years: 2019-2021 Sample size: It will include all patients presented to our department fulfilling the inclusion criteria.

Study population: The study will be conducted in patients with Incompetent Great saphenous vein

Inclusion criteria:

• Primary symptomatic VVS (CEAP, C3eC6), sapheno-femoral junction (SFJ) incompetence, GSV reflux from the groin to below the knee

Exclusion criteria:

• Exclusion criteria included a history of venous surgery, suspected or proven deep venous thrombosis, reflux of deep veins to distal limb, duplication of GSV, and patients' refusal to participate in the trial.

Consent: Patients after signing informed consent that possible complication from the procedure ought to happen and what are the alternatives.

Data collection: The demographics, Symptoms and preoperative clinical data will be collected History Data: included patient's demographics, underlying medical conditions, any previous associated morbidity.

Examination: Venous examinations. Laboratory: Blood picture, Blood sugar level, Kidney functions, Liver functions and Coagulation profile.

Imaging: Duplex US Method of Randomization: Computer based Therapies Surgical group. Conventional surgical procedures will carried out through a 3-4 cm incision in the groin. The trunk of GSV and the tributaries will be ligated and divided. The GSV will be removed using a pin-stripper, and all varices and incompetent perforators will be removed by phlebectomy.

Microwave group. The microwave treating wire (Microwave Intracavity Coagulation System; Shanghai Medical Electronics, Shanghai, China) will be inserted into the GSV until it reached the medial aspect of ankle, guided by a light that illuminated the tip of the wire. Then, GSV will be ablated using pulse mode at 20-30 W. The treating wire will be withdrawn at 2-4 mm/s, with the ablation time lasting 2 s (energy delivery to the GSV was estimated at around 80 J/cm); the treatment parameters will be based on a previous report. Tumescence will be used in all patients with 0.9% saline containing 20 mL 2% lidocaine with 1: 200,000 adrenaline and 20 mL 0.5% levobupivacaine in 1 L 0.9% saline.

Laser ablation group: Endovenous Laser Ablation (EVLA) uses a laser Fiber, which is inserted into the abnormal vein via a small skin puncture.using 1470 nm laser and a "radial" fiber for less discomfort. Two weeks later the "branch vessels" have reduced in size Radiofrequency ablation group: inserts a small catheter into the diseased vein through a small incision, using ultrasound guidance for an accurate and live view. Consistent and uniform heat is delivered to contract the collagen in the vein walls, causing them to collapse and close. After the vein is closed the treated vein is gradually absorbed into surrounding tissue

Follow up

Criteria for technical success will be:

1. Closed or absent GSV with lack of flow
2. A re-canalized GSV or treatment failure will be defined as an open segment of the treated vein segment of >10 cm in length.
3. All patients will be followed as outpatients up at 1, 3, 6, 12, and 24 months after surgery.
4. The operation time, number of incisions, intraoperative blood loss (determined by the swabs weighed pre and postoperatively)
5. Recurrence of varicosities will be recorded, as well as any complications.

The criteria for assessment:

1. Ecchymosis was confirmed 72 h after operation when the lividity and congestion area was >1 cm2 in the affected limbs.
2. Skin burns were identified 72 h after operation when the skin was red and oedematous according to the criteria for burns.
3. Recurrence was defined by both duplex ultrasound and the clinical examination. A varicose vein that had not been observed before or previously been marked by the patient on the AVVQ form was considered to be a recurrent varicose vein (owing to neo-vascularization or dilation of pre-existing veins).
4. Sensory impairment (numbness) that occurred around incisions was recorded based on the patient's history and physical examination.

QoL assessment The diseased relation effect on QoL was determined using the AVVQ (Chinese version), which assessed the specific effect on QoL and was scored from 0 (no effect of VVS on QoL) to a theoretical maximum of 100.8 The VCSS (Chinese version) was also completed (for the VCSS, 0 represents no significant venous disease and 30 is the maximum score), which is a valid sensitive and responsive measure of the severity of VVS.

ELIGIBILITY:
Inclusion Criteria:

* Primary symptomatic VVS (CEAP, C3 , C6),
* Sapheno-femoral junction (SFJ) incompetence, GSV reflux from the groin to below the knee

Exclusion Criteria:

* A history of venous surgery, suspected or proven deep venous thrombosis,
* Reflux of deep veins to distal limb
* Duplication of GSV
* Patients' refusal to participate in the trial.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-06-18 (Actual); Primary Completion 2021-06-18 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
Great Saphenous vein patency | 6 months
  Lack of flow or closed great saphenous vein
Operation Time | intraoperative
  The time of the whole procedure

SECONDARY OUTCOMES:
Recurrence varicose vein | 12 Months
  varicose veins reappear again after the operation
Adverse effect of the procedure | 12 Months
  Thrombophlebitis, infection or blood loss

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Mansoura, Al Mansurah, Mansoura University
  - Mansoura University Hospital, Al Mansurah

IPD SHARING:
Plan to Share IPD: No